CLINICAL TRIAL: NCT00515658
Title: Antidepressant Effect of Theta-Burst rTMS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Rambam2141_CTIL
Record Dates: First submitted 2007-08-13; First posted 2007-08-14 (Estimated); Last update posted 2007-08-14 (Estimated); Status verified 2007-08

CONDITIONS: Major Depression
Keywords: Major depression; Theta-burst rTMS; Cortical excitability; Hamilton depression rating scale
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: theta-burst rTMS

SUMMARY:
The aim of this study is to evaluate the safety and efficacy of theta-burst rTMS in patients with major depression. Patients will be randomized to receive ether left-sided intermittent theta-burst rTMS or rigt-sided continuous theta-burst rTMS or sham theta-burst rTMS over two weeks period with an option for an additional two weeks period, depending on treatment response. Clinical assessments will be performed weekly by the Hamilton depression rating scale. In addition, standard neurophysiological assessment of cortical excitability will be done.

ELIGIBILITY:
Inclusion Criteria:

* Major depressive episode (DSM IV criteria).
* Informed consent.
* Age: 18-70.

Exclusion Criteria:

* Suicidality
* Psychosis
* Pacemaker
* Cardiac arrythmia
* seizure disorder
* implantable metal devices
* PNS and CNS disorders
* any other contraindications as specified in safety guidelines for rTMS (Wassermenn, 1998).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2007-03

CONTACTS AND LOCATIONS:
Overall Officials: Ehud Klein, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Medical Center, Haifa, Israel